CLINICAL TRIAL: NCT04362423
Title: A Pilot Study to Evaluate Functional Near Infrared Spectroscopy to Detect Pain in Infants and Young Children Under General Anesthesia
Brief Title: Functional Near Infrared Spectroscopy to Detect Pain in Young Children Under General Anesthesia
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-3578
Record Dates: First submitted 2015-08-12; First posted 2020-04-27 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Pain
Keywords: Acute pain measurement in children
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- propofol+fNIRS: During data collection, only propofol is used to maintain the anesthesia. Peripheral noxious stimuli produced from the neurophysiological monitoring (SSEP)
  Interventions: Device: fNIRS
- sevoflurane+fNIRS: During data collection, only sevoflurane is used to maintain the anesthesia. Peripheral noxious stimuli produced from the neurophysiological monitoring (SSEP)
  Interventions: Device: fNIRS
- neuro-stimulator+fNIRS: During data collection, we use neuro-stimulator to give the stimulation.
  Interventions: Device: fNIRS

INTERVENTIONS:
Device: fNIRS — Near infrared spectroscopy (NIRS) is a non-invasive, portable, relatively inexpensive optical technology similar to pulse oximetry except that it measures total hemoglobin, oxy-hemoglobin, and deoxyhemoglobin in brain tissue (capillaries) rather than arteries.
  Other Names: Functional Near Infrared Spectroscopy

SUMMARY:
This is a three-phase pilot prospective study to develop a devise capable of detecting changes in cortical blood volume and oxygenation due to noxious stimuli. The hypothesis of the study is that optical signal changes corresponding to blood volume and oxygenation will be detected with functional near infrared spectroscopy in the prefrontal cortex of children under general anesthesia in response to peripheral noxious stimuli produced from the neurophysiological monitoring (SSEP).

DETAILED DESCRIPTION:
Pain is a subjective feeling, and an objective measure of pain is needed to obtain improved clinical management and safe outcomes of pain treatment. At present, there is a lack of specific physiological markers of acute pain that can guide analgesic treatment both during and after surgery. The anesthesiologist typically relies on hemodynamic variables to guide administration of opioids for surgical pain, but those parameters are not always either specific or sensitive. On the other hand, uncontrolled pain during surgery can lead to emotional distress and enhancement of the systemic inflammatory response (1).

Current evidence (2-4) shows that the prefrontal cortex plays an important role in pain perception and emotional elaboration. Functional neuroimaging (functional magnetic resonance imaging functional magnetic resonance imaging (fMRI) functional near infrared spectroscopy fNIRS) has been recently utilized to investigate cerebral pain-related activity (5, 6).

The investigators propose to detect the optical signal changes over the prefrontal cortex using fNIRS and diffuse optical imaging (DOI) in response to noxious electrical stimulation. This electrical stimulation will be applied over the ulnar nerve at the wrist in children undergoing neurosurgery with SSEP monitoring. This noxious electrical stimulation is the standard stimulus used to establish baseline somatosensory evoked potentials in this patient population for this surgery. DOI is a mathematical methodology used to generate an image from the optical signals analogous to the mathematical methodology of generating a MRI from nuclear magnetic spectroscopy signals.

The investigators will evaluate the magnitude of change of fNIRS-DOI signals after two different intensities of noxious electrical stimulation and following intravenous administration of fentanyl (2 mcg/kg). The investigators will also analyze the temporal correlation of the prefrontal cortex fNIRS-DOI changes with the SSEPs. The results will lead to the identification of an objective specific biomarker for acute pain in children. Our long-term goal is to develop a portable and readily accessible device to improve management of intraoperative nociception and to evaluate acute pain in awake non-verbal children.

ELIGIBILITY:
Inclusion Criteria:

* They are presenting for tethered spinal cord release , posterior fossa decompression, or spine surgery;
* They are between 1 month to 16 years of age;
* Their anesthetic plan includes endotracheal intubation and neuromonitoring;

Exclusion Criteria:

* Patients with a known history of chronic pain;
* Patients with abnormal frontal lobe brain structure or abnormality of forehead precluding the fNIRS probe securement;
* Patients with a known allergy to fentanyl;
* Patients with unstable hemodynamics.
* Patients with a contraindication to the use of propofol

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The patients who are presenting to CCHMC for tethered spinal cord release , posterior fossa decompression, or spine surgery; the anesthetic plan includes endotracheal intubation and neuromonitoring.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
the changes of oxy-, deoxy-, total-hemoglobin | during stimulation (16 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Yifei Jiang, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States